CLINICAL TRIAL: NCT04056988
Title: Utilizing Contrast-enhanced Ultrasound (CEUS) to Assess Critically Hypo Perfused Spinal Cord Tissue After Injury
Brief Title: tSCI Contrast Enhanced Ultrasound Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Christoph Hofstetter, Assistant Professor, School of Medicine: Neurological Surgery, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00003267
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Acute Spinal Cord Injury
MeSH Terms: interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Acute spinal cord injury patients to undergo contrast-enhanced (Experimental): Perflutren lipid microsphere preparation is an ultrasound contrast agent. Ultrasound contrast agents are used to help provide a clear picture during ultrasound.
  A hand-held intraoperative ultrasound probe will be used to collect sagittal images of the spinal cord centered above the spinal cord injury. A bolus IV injection of DEFINITY® contrast agent (1.5ml DEFINITY®/8.5ml saline) will be given. Continuous imaging will be obtained to record contrast inflow and washout.
  Interventions: Drug: Perflutren Lipid Microsphere

INTERVENTIONS:
Drug: Perflutren Lipid Microsphere — Perflutren lipid microsphere preparation is an ultrasound contrast agent. Ultrasound contrast agents are used to help provide a clear picture during ultrasound.
  Other Names: DEFINITY®

SUMMARY:
Patients with traumatic spinal cord injury (tSCI) often suffer from spinal cord swelling inside the thecal sac, which contains the spinal cord and surrounding fluid, leading to increased pressure on the spinal cord tissue and decreased spinal cord blood flow at the site of injury. The combination of increased pressure and decreased blood flow causes vascular hypo-perfusion of the spinal cord and exacerbates the severity of the injury. This is also referred to as secondary injury. Thus, knowledge of spinal cord hypo-perfusion would allow the treating physician to optimize the hemodynamic condition of patients with acute spinal cord injury and potentially improve functional outcomes. The investigators plan to use contrast-enhanced ultrasound (CEUS) to determine the decrease of blood flow in the spinal cord at the site of injury, during the routine surgery that these patients require to decompress and stabilize their injured spine. This may help the investigators to determine the efficacy of certain treatments in improving blood flow and patients suffering from tSCI.

DETAILED DESCRIPTION:
Patients presenting to the Harborview Emergency Room with acute traumatic spinal cord injury (tSCI) will be recruited to undergo contrast-enhanced ultrasound (CEUS) during routine surgery for decompression and stabilization of their injury.

Traumatic spinal cord injury (tSCI) develops in two phases. The primary injury is characterized by direct mechanical destruction of cells, nerve fibers, and blood vessels. The secondary injury phase represents the downstream biological effects of the loss of blood flow in the injury center as well as significant hypoperfusion in the surrounding penumbral zone. This process is associated with cytotoxic spinal cord edema, which causes a rise in tissue pressure within the contused spinal cord. While experimental studies demonstrate that spinal cord tissue damage due to primary injury is often remarkably limited, the cascade of biochemical and molecular processes that comprise secondary injury often exacerbate and define the extent of injury to the patient.

Accordingly, two routinely performed clinical treatment strategies aim to mitigate the effects of secondary injury by improving the local tissue perfusion of the contused spinal cord. First, surgical decompression of the spinal cord is recommended within 24 hours after injury, as it may improve functional outcomes. Second, trauma guidelines recommend the maintenance of the mean arterial blood pressure at 85 - 90 Hg for the first 7 days after acute spinal cord injury.

Despite these interventions and a tremendous research effort to develop neuroprotective therapies targeting the hypoperfused "rescue-able" penumbral zone, there are no clinically efficacious techniques to improve functional outcomes following tSCI. The investigators believe that a lack of clinical biomarkers for the hypoperfused "rescue-able" penumbral zone is the main roadblock to the development of novel therapeutic procedures and therapies. This motivates a search for a biomarker for tSCI that can guide surgical and critical care interventions. The investigators seek to develop an ultrasound-based biomarker for tSCI that is sensitive to the underlying tissue pathology and predictive of clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* >18
* Male or Female
* Acute <72 hours spinal cord injury (ASIA) grade A to D
* Medically stable to undergo routine decompression and spinal realignment

Exclusion Criteria:

* <18 years of age
* Not clinically stable for spinal surgery
* Traumatic Brain Injury
* Known sensitivity to lipid microsphere or its components i.e., (PEG).
* A history of anaphylactoid reactions from ultrasound-enhancing agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Use of CEUS to improve post operative outcomes in acute spinal cord injury | Intra-operative
  Contrast-enhanced ultrasound (CEUS) to determine decrease of blood flow in the spinal cord at the site of injury

CONTACTS AND LOCATIONS:
Overall Officials: Christoph P Hofstetter, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States